CLINICAL TRIAL: NCT00324779
Title: Multicenter Therapy Study for Children With Mature B-NHL or B-ALL With a Rituximab - Window Before Chemotherapy
Brief Title: Rituximab in Treating Young Patients Who Are Receiving Chemotherapy for B-Cell Non-Hodgkin's Lymphoma or B-Cell Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Erlangen (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000466643; B-NHL-BFM-Rituximab; EU-205119; NHL-BFM-RITUXIMAB
Record Dates: First submitted 2006-05-10; First posted 2006-05-11 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Leukemia; Lymphoma
Keywords: B-cell childhood acute lymphoblastic leukemia; untreated childhood acute lymphoblastic leukemia; stage I childhood large cell lymphoma; stage II childhood large cell lymphoma; stage III childhood large cell lymphoma; stage IV childhood large cell lymphoma; stage I childhood lymphoblastic lymphoma; stage II childhood lymphoblastic lymphoma; stage III childhood lymphoblastic lymphoma; stage IV childhood lymphoblastic lymphoma; stage I childhood small noncleaved cell lymphoma; stage II childhood small noncleaved cell lymphoma; stage III childhood small noncleaved cell lymphoma; stage IV childhood small noncleaved cell lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Burkitt Lymphoma | interventions — Rituximab

INTERVENTIONS:
Biological: rituximab

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some find cancer cells and kill them or carry cancer-killing substances to them. Others interfere with the ability of cancer cells to grow and spread. Giving rituximab before chemotherapy may be an effective treatment for B-cell non-Hodgkin's lymphoma or B-cell acute lymphoblastic leukemia.

PURPOSE: This phase II trial is studying how well rituximab works in treating young patients who are planning to receive chemotherapy for B-cell non-Hodgkin's lymphoma or B-cell acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate in children and adolescents with B-cell non-Hodgkin's lymphoma (B-NHL) or B-cell acute lymphoblastic leukemia (B-ALL) treated with rituximab monotherapy as upfront window therapy before chemotherapy.
* Evaluate the effect of rituximab on different histological subtypes of childhood mature B-NHL or B-ALL in patients treated with this regimen.
* Investigate the rituximab response in patients treated with this regimen.
* Determine the toxicity profile of rituximab in these patients.
* Collect pharmacokinetic and pharmacodynamic data from patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive rituximab IV on day 1.

PROJECTED ACCRUAL: A total of 79 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically and immunohistochemically OR cytomorphologically and immunphenotypically confirmed mature B-cell non-Hodgkin's lymphoma or B-cell acute lymphoblastic leukemia
* CD20 positive disease

PATIENT CHARACTERISTICS:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* Adequate general condition with sufficient organ function (hepatic, renal, and cardiac)
* No known disease that would preclude protocol therapy with rituximab
* No known allergies against proteins
* No acute or previous hepatitis B infection

PRIOR CONCURRENT THERAPY:

* At least 2 weeks since prior corticosteroids
* No prior radiotherapy
* No prior or concurrent chemotherapy
* No concurrent treatment in another investigational trial

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 79 (Estimated)
Dates: Start 2004-03; Primary Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Response rate
Effect of rituximab on different histological subtypes
Rituximab response
Toxicity
Pharmacokinetics and pharmacodynamics

CONTACTS AND LOCATIONS:
Overall Officials: Alfred Reiter, MD, Study Chair — University Hospital Erlangen
Locations (38):
- Germany (37):
  - Kinderklinik - Universitaetsklinikum Aachen, Aachen
  - Klinikum Augsburg, Augsburg
  - Charite - Campus Charite Mitte, Berlin
  - Helios Klinikum Berlin, Berlin
  - Evangelisches Krankenhauus Bielfeld, Biefeld
  - Klinikum Bremen-Mitte, Bremen
  - Children's Hospital, Cologne
  - Vestische Kinderklinik, Datteln
  - Universitatsklinikum Carl Gustav Carus, Dresden
  - Helios Klinikum Erfurt, Erfurt
  - Universitaets - Kinderklinik, Erlangen
  - Universitaetsklinikum Essen, Essen
  - Klinikum der J.W. Goethe Universitaet, Frankfurt
  - Universitaetskinderklinik - Universitaetsklinikum Freiburg, Freiburg im Breisgau
  - Kinderklinik, Giessen
  - Klinik und Poliklinik Fuer Kinder-und Jugendmedizin - Universitaetsklinikum Greifswald, Greifswald
  - University Medical Center Hamburg - Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitaets-Kinderklinik Heidelberg, Heidelberg
  - Universitaetsklinikum des Saarlandes, Homburg
  - Universitaets - Kinderklinik, Jena
  - Staedtisches Klinikum Karlsruhe gGmbH, Karlsruhe
  - Kinderkrankenhaus Park Schoenfeld, Kassel
  - University Hospital Schleswig-Holstein - Kiel Campus, Kiel
  - Universitaets - Kinderklinik, Leipzig
  - Universitaets - Kinderklinik - Luebeck, Lübeck
  - Universitatsklinikum der MA, Magdeburg
  - Universitaets - Kinderklinik, Marburg
  - Krankenhaus Muenchen Schwabing, Munich
  - Dr. von Haunersches Kinderspital der Universitaet Muenchen, Munich
  - Klinik und Poliklinik fuer Kinder und Jugendmedizin - Universitaetsklinikum Muenster, Münster
  - Cnopf'sche Kinderklinik, Nuremberg
  - Klinik St. Hedwig-Kinderklinik, Regensburg
  - Olgahospital, Stuttgart
  - Universitaetsklinikum Tuebingen, Tübingen
  - Comprehensive Cancer Center Ulm at Universitaetsklinikum Ulm, Ulm
  - Universitaets - Kinderklinik Wuerzburg, Würzburg
- University Children's Hospital, Zurich, Switzerland